CLINICAL TRIAL: NCT03659110
Title: Post-Approval Safety Monitoring Program to Assess the Safety Profile of GARDASIL in China Usual Practice
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Chaoyang District Centre for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Other Study IDs: cycdc2018-1
Record Dates: First submitted 2018-09-03; First posted 2018-09-06 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Cervical Cancer
Keywords: vaccine; safety
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1000 subjects receive the HPV 4 vaccine
  Interventions: Biological: HPV 4

INTERVENTIONS:
Biological: HPV 4 — 1000 subjects will be received the HPV 4 vaccine

SUMMARY:
This is a post-Approval Safety Monitoring Program to assess the safety profile of GARDASIL in china usual practice.

ELIGIBILITY:
Inclusion Criteria:

* Any person who is intended to be inoculated with first dose GARDASIL based on his/her own wishes at screening

Exclusion Criteria:

1. Unable to provide written informed consent
2. Any woman who is known being pregnant at screening
3. Subject who is participating or going to participate in another study which involves GARDASIL administration

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Volunteers aged 20-45 years
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the Rate of Adverse reactions of GARDASIL in China usual practice | 24 months
  Adverse reactions associated with vaccine will be observed in females Aged 20-45 Years after vaccination. Solicited local adverse events include Pain, Redness, Swelling, Induration, Rash, Pruritus at injection site. solicited general adverse events include Fever, Nausea, Vomiting, Diarrhea, Decreased appetite, Be agitated (irritability, abnormal crying), fatigue, allergy
Number of participants with adverse events following any dose of vaccine | within 30 days after each dose
  Number of participants with adverse events following any dose of vaccine